CLINICAL TRIAL: NCT03375879
Title: The Role of Bandage Contact Lens in Post-operative Patients Undergoing Fasanella Servat Ptosis Repair
Brief Title: Bandage Contact Lens in Post Operative Ptosis Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: St. Joseph's Healthcare Hamilton (Other)
Collaborators: Robert Adam (Unknown); Forough Farrokhyar (Unknown); Sivisan Suntheralingam (Unknown)
Responsible Party: Principal Investigator, John Harvey, Director of Oculoplastic, Reconstructive, Lacrimal and Orbital Service, St. Joseph's Healthcare Hamilton
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: StJosephharveyj
Record Dates: First submitted 2017-11-08; First posted 2017-12-18 (Actual); Last update posted 2018-04-23 (Actual); Status verified 2018-04

CONDITIONS: Ptosis; Blepharoptosis
Keywords: Ptosis; Blepharoptosis; bandage contact lens; fasanella servat procedure
MeSH Terms: conditions — Blepharoptosis

STUDY DESIGN:
Intervention Model Description: The investigators will place a contact lens on both eyes and immediately take it off from one (this will be the sham lens eye). Randomization of the lens placement will be determined by a flip of a coin (heads - keep lens on right eye. Tails - keep lens on left eye). Investigator will randomly generate for each patient whether the contact lens will be kept on right or left eye, sham contact lens will be placed on other eye, placing it and immediately removing it. Therefore, the patient will not know which eye has a lens.
Who Masked: Participant
Masking Description: The investigator will place a contact lens on both eyes and immediately take it off from one (this will be the sham lens eye). Randomization of the lens placement will be determined by a flip of a coin (heads - keep lens on right eye. Tails - keep lens on left eye). Investigator will randomly generate for each patient whether the contact lens will be kept on right or left eye, sham contact lens will be placed on other eye, placing it and immediately removing it. Therefore, the patient will not know which eye has a lens.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Bandage contact lens (Active Comparator): Placing a bandage contact lens in one eye.
  Interventions: Device: Bandage contact lens
- Sham contact lens (immediate removal) (No Intervention): Sham contact lens will be placed on other eye, placing it and immediately removing it so patient does not know which eye will have a bandage contact lens.

INTERVENTIONS:
Device: Bandage contact lens — Bandage contact lens
  Arms: Bandage contact lens

SUMMARY:
This study is being conducted to determine whether the use of bandage contact lens after ptosis surgery provides any benefits for the patient or is unnecessary.

DETAILED DESCRIPTION:
This study is being conducted to determine whether the use of bandage contact lens after ptosis surgery provides any benefits for the patient or is unnecessary. The investigators hope to show through questionnaires based on the patient's experience after their surgery to see if the bandage contact lens has provided any benefit for the patient. This is a randomized control trial in which patients undergoing bilateral ptosis surgery (Fasanella servat procedure) will have one of their eyes randomized to receive a bandage contact lens after surgery while the other eye will not receive anything.In this randomized control trial, patients requiring surgery with bilateral ptosis will have one eye randomized to receive a bandage contact lens whereas the other eye will not after their surgery. Follow up will occur in one week where the outcomes will be obtained through questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* patients who have bilateral ptosis (drooping eyelids) and will require surgery to correct this

Exclusion Criteria:

* patient having any other eye related pathologies

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2018-02-21 (Actual); Primary Completion 2018-12-01 (Estimated); Study Completion 2018-12-01 (Estimated)

PRIMARY OUTCOMES:
Patient's pain/discomfort | One week post-operation.
  This will be obtained using the Eye Sensations Scale where the patient can select a box from None, Mild, Moderate, Severe, to Extreme.

SECONDARY OUTCOMES:
Blurry vision | One week post-operation.
  This will be measured using one question from the Ocular Surface Disease Index (OSDI), with a scale from 0 (none of the time) to 4 (all of the time).

CONTACTS AND LOCATIONS:
Locations (1):
- St. Joseph's Hospital Hamilton, Hamilton, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No
IPD will not be shared with others.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-10-17): https://cdn.clinicaltrials.gov/large-docs/79/NCT03375879/Prot_SAP_000.pdf